CLINICAL TRIAL: NCT04395131
Title: Clearum High Flux Hemodialyzer: Safety and Performance Clinical Study
Brief Title: Clearum High Flux Hemodialyzer Used in Hemodialysis for Subjects With End-Stage Renal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SA0720191
Record Dates: First submitted 2020-04-30; First posted 2020-05-20 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: End-stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clearum HF Dialysis Subjects (Other): All subjects enrolled in the study and treated with the Clearum HF hemodialyzer
  Interventions: Device: Clearum HF Hemodialyzer

INTERVENTIONS:
Device: Clearum HF Hemodialyzer — the hemodialyzer will be used 3x week for 3.5-4.5 hours with a Qb of at least 350 ml/min

SUMMARY:
The study will be a prospective, interventional, non-randomized, single-center study in 20 ESRD patients on hemodialysis. The study will compare performance of the Clearum HS dialyzer to typical values obtained with other commercially available high flux dialyzers. In addition, the Clearum HS dialyzer will be compared to a Fresenius FX80 dialyzer for a baseline (control) comparison. This will be a post-market study. The duration of the trial is 2 weeks for the FX80 control dialyzer + 6 weeks with the Clearum HS dialyzer used for 3x weekly high flux hemodialysis.

DETAILED DESCRIPTION:
The study will compare performance to typical values obtained with commercially available dialyzers used for high flux hemodialysis and comparing the Clearum HS dialyzer to the baseline values of a control FX80 Dialyzer.

The duration of the trial is 2 weeks for the FX80 control dialyzer + 6 weeks with the Clearum HS dialyzer used for 3x weekly high flux hemodialysis.

The sampling, reported in Table 1 below, will be done at mid-week sessions (pre and post session sampling) and consists of a blood draw for baseline dialysis with the FX80 weeks 1 and 2, or Clearum HS dialyzer at weeks 3, 5 and 8 for uremic toxins: urea, creatinine, phosphate, B2-microglobulin, albumin, sodium, potassium, calcium, magnesium, platelets and leucocytes, and platelets. In addition, a presession sample will be taken for coagulation parameter TAT, hematocrit and inflammatory markers IL6 and C reactive protein at baseline for FX80 at mid-week sessions during weeks 1 and 2 and during weeks 3, 5 and 8 for the Clearum HS dialyzer.

Instantaneous B2M clearance sampling will be done at week 7 during the Clearum HS dialyzer phase and consists of a blood sample prior to the dialyzer and immediately after the dialyzer at two time points, 15-30 min and at 120-150 min, respectively.

Blood rest will be done by comparing the dialyzer to a set of 5 illustrations and giving a score of 1 (worst) to 5 (best) that best correlates the dialyzer with the illustration, at the end of the dialysis session after blood has been returned to the patients (both FX80 and Clearum HS) on the sampling days.

The patients will be treated for 2 weeks with a standard dialyzer (FX80) and an additional 6 weeks with the Clearum HS dialyzer (experimental period). Both hemodialyzers will be used for 3 times a week. Expected duration for the study including enrolment will be 3 months.

The study duration will be approximately 3-4 months. Each patient will receive 6 hemodialysis sessions with FX80 and 18 sessions with Clearum HS hemodialyzer, and the treatment time will be between 3.5 and 4.5 hours

ELIGIBILITY:
Inclusion Criteria:

* ESRD Patients aged 18 years or older
* Patients able to give informed consent (IC) and interested to participate in the study
* Stable (according to the investigator) on hemodialysis for more than 3 months with previous treatments of 3x weekly hemodialysis or hemodiafiltration
* Stable hemoglobin between 10 and 12 g/dl in the most recent two consecutive blood draws
* Stable anticoagulation and ESA regimen with no dosing modifications in the past 1 month
* Patients who have an adequate AVF or graft, capable of providing a blood flow rate of at least 300 mL/min according to sessions conducted in past month

Exclusion Criteria:

* Patients who have acute renal failure with the chance for recovery.
* Patients who are pre-scheduled for a living kidney transplant within the next two months, who plan a change to PD within the next two months or who require single needle dialysis therapy.
* Pregnant and lactating women.
* Patients with a history of positive serology tests for Hepatitis B surface antigen, positive Hepatitis C total antibody, HIV and syphilis.
* Patients with known hemodynamic instability, anemia (Hgb < 90 g/L), and/or severe bleeding risks secondary to coagulation disorders.
* Patients with active or ongoing infection per investigator's judgement.
* Patients with a history of solid tumors requiring anti-cancer therapy in the past or next 6 months or a life expectancy less than 1 year or patients with a history of a hematology neoplasm.
* Patients diagnosed with a NYHA Class IV congestive heart failure, or acute coronary syndrome and/or who have suffered a myocardial infarction within three months prior to the start of the study.
* Patients with a history of severe mental disorders.
* Patients who are currently participating or have previously participated in another interventional clinical trial in the past 4 weeks.
* Patients who have had an allergic response to polyarylethersulfone (PAES) or polysulfone membranes or have a history of poor tolerance to dialyzers with synthetic membranes.
* Patients with advanced liver, heart or pulmonary disease as judged by the Investigator
* Patients with any comorbidity possibly conflicting with the study purpose or procedures as judged by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
Evaluate performance of small-solute (toxin) removal | End of dialysis treatment
  The primary objective of this study is to evaluate performance of small-solute (toxin) removal, represented by urea, under standard high flux hemodialysis conditions with a mean urea reduction ratio (URR) of 65% or greater.

SECONDARY OUTCOMES:
Adverse Events | 8 weeks, 3 sessions per week
  Evaluate of all adverse events during the study period
B2M reduction ratio | 5 sampling at mid-week session of week 1, 2, 3, 5 and 8
  Evaluate performance of the B2M reduction ratio
Instantaneous clearance of B2M during specified time-points | 1 sampling at mid-week session of week 7
  Evaluate the instantaneous clearance of B2M for the Clearum HS dialyzer at 15-30 min and at 120-150 min at session the mid-week session of week 2 with the Clearum dialyzer.
Reduction ratio of albumin during hemodialysis | 5 sampling at mid-week session of week 1, 2, 3, 5 and 8
  Evaluate the reduction ratio of albumin during the hemodialysis session with the Clearum dialyzer and any trends in albumin concentration over a 6-week period
Follow-up of CRP for patients treated with Clearum dialyzer | Kinetic over 6 week period
  Observe the trends in inflammatory markers CRP over a 6-week period
Follow-up of IL6 for patients treated with Clearum dialyzer | Kinetic over 6 week period
  Observe the trends in inflammatory markers IL6 over a 6-week period
Evaluation of TAT (Thrombin-antithrombin) complex | End of dialysis treatment
  Evaluate coagulation parameters as assessed by Thrombin-anti-thrombin (TAT) on the dialyzer after blood restitution at the end of the dialytic session for sessions where sampling occurs
Quality of rinse-back (filter and circuit) via a visual scale | End of dialysis treatment
  Evaluate on a qualitative photo visual score ranging from poor to very good (1-5) for the residual blood remaining in the dialyzer after rinse back at the end of the session

CONTACTS AND LOCATIONS:
Locations (1):
- DaVita Clinical Research Germany, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No